CLINICAL TRIAL: NCT05170464
Title: Comparing the Acute Effects of Exercise and Caffeine on Working Memory During a Short Period of Caffeine Deprivation in Moderate to Heavy Caffeine Consumers
Brief Title: The Acute Effects of Exercise and Caffeine on Working Memory During Acute Caffeine Deprivation
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Western University, Canada (Other)
Responsible Party: Principal Investigator, Dr. Harry Prapavessis, Professor, School of Kinesiology, Western University, Canada
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 120038
Record Dates: First submitted 2021-12-10; First posted 2021-12-28 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-02

CONDITIONS: Acute Exercise; Caffeine Withdrawal; Memory Deficits
MeSH Terms: conditions — Memory Disorders | interventions — Exercise

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Acute Exercise (Experimental): 20 minutes of moderate intensity acute exercise (treadmill speed to achieve ⅔ of maximum heart rate).
  Interventions: Behavioral: Acute Exercise
- Caffeine Ingestion (Active Comparator): 1.2mg/kg of powdered caffeine (Caffeine powder, ReagentPlus® from Sigma-Aldrich) dissolved in 1 cup of water then sitting for 20 minutes.
  Interventions: Drug: Caffeine Powder

INTERVENTIONS:
Behavioral: Acute Exercise — Brisk walking on a treadmill at ⅔ maximum heart rate as defined by 220-age (in years).
  Other Names: Aerobic Exercise
  Arms: Acute Exercise
Drug: Caffeine Powder — Participants will receive powdered caffeine dissolved in one cup of water (1.2mg/kg)
  Other Names: Caffeine Ingestion
  Arms: Caffeine Ingestion

SUMMARY:
To determine the effects of moderate intensity exercise and caffeine on working memory in deprived caffeine consumers.

DETAILED DESCRIPTION:
Participants will be asked to keep consumption of caffeine before the first visit to their regular dose (ex. morning coffee) and to abstain from alcohol and drugs for at least 18 hours prior to testing. Participants will be urged to arrive at the same time for each visit. Upon arrival to the Exercise and Health Psychology lab (located in room 408 of the Arthur and Sonia Labatt Health Science Building at Western University) participants will be given the letter of information and asked to sign the informed consent form. Participants will also be asked to complete a demographic survey, PAR-Q (Physical Activity Readiness Questionnaire) readiness for exercise, Godin Leisure-Time Exercise Questionnaire, CCQ-R (Caffeine Consumption Questionnaire), and the CWSQ (Caffeine Withdrawal Symptom Questionnaire). Vitals (heart rate and blood pressure) will be assessed following the completion of the questionnaires as well as post assessment in the seated position. Prior to evaluation on the N-back task (cognitive memory task described below) a practice stage with be conducted until the participant can consistently score 75% or higher on three consecutive trials to eliminate a learning effect. After establishing familiarity, a baseline cognition score will be conducted through the n-back assessment.

Prior to arrival for the second visit, participants will be asked to refrain from caffeine for at least 24 hours and to abstain from abstain from alcohol and drugs for at least 18 hours prior to testing. During the second visit (approximately 24 hours after the first) the participants will complete the pre-caffeine or pre-exercise questionnaire, the CWSQ and vitals will be monitored pre and post intervention. Caffeine abstinence will be validated through self-report with the use of deception (participants being told that their saliva sample is being tested for the presence of caffeine). To collect saliva, a cotton swab will be placed under their tongue for 1minute, placed into a tube, and then a co-investigator will discard the tube into a biohazard deposal container immediately. Participants will then complete another n-back assessment.

The participants will be randomized into either the moderate intensity exercise or caffeine ingestion group. The interventions are as followed; Moderate Intensity Exercise will consist of a 20-minute bout of moderate intensity aerobic exercise. Exercise will consist of a 2-minute warm-up, followed by 15 minutes of walking at a rate, which will allow you to reach 2/3 of your max heart rate (moderate intensity exercise= (220-age) x 0.6), and then a 3-minute cool down on a treadmill (together equaling 20 minutes). HR will be monitored through heart rate monitors worn by the participants. The caffeine ingestion group will ingest 1.2 mg/kg of caffeine in powder form with water to drink, after ingestion of caffeine participants will wait 20 minutes to ensure peak plasma levels. The post intervention n-back assessment will begin within two minutes of the completion of either intervention.

ELIGIBILITY:
Inclusion Criteria:

* Are over the age of 18 years
* Consume at least 150 mg of caffeine a day
* Do not have any cognitive problems
* Are not pregnant
* Do not have a medical condition that prevents you to exercise
* Do not have an orthopaedic limitation
* Have access to a telephone or an email account for communication
* Can read and write in English

Exclusion Criteria:

* Participants taking prescription medication for depression or anxiety
* Participants that cannot give informed consent will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2022-01-10 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Change in Working Memory as assessed by N-back task | Baseline and 24 hours later (deprived and post-treatment).
  Participants will complete three n-back assessments, one baseline, one after 24 hours of caffeine deprivation, and one after treatment (either caffeine ingestion or acute exercise). Percent error rates will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Harry Prapavessis, PhD, Principal Investigator — Western University
Locations (1):
- The University of Western Ontario, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided
Given the lack of research currently, it is unlikely for other researchers to request data. If other studies are done, we will put together a plan to share IPD.

REFERENCES:
- [Background] Morava A, Fagan MJ, Prapavessis H. Effects of Caffeine and Acute Aerobic Exercise on Working Memory and Caffeine Withdrawal. Sci Rep. 2019 Dec 23;9(1):19644. doi: 10.1038/s41598-019-56251-y. PMID 31873185